CLINICAL TRIAL: NCT05714436
Title: Understanding and Identifying Priorities for Improving the Healthcare Experiences of People With Incurable Head and Neck Cancer: a Qualitative Investigation and Co-design Approach
Brief Title: Ii-HANC Improving Incurable Head and Neck Cancer Healthcare Experiences
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); University of Newcastle Upon-Tyne (Other); University of Liverpool (Other); Lancaster University (Other)
Responsible Party: Sponsor
Other Study IDs: STH21983
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Work Package 1a: Longitudinal interviews with patients and family carers to generate thematic framework for co-design workshops
- Work Package 1b: On-line focus groups with healthcare professionals to generate thematic framework for co-design workshops
- Work Package 2: Co-design workshops to generate decisions about priority areas for intervention development

SUMMARY:
This research aims to improve experiences of patients with incurable head and neck cancer (IHNC) by finding out the most pressing issues for them and developing solutions to improve these.

Patients with IHNC have many complex needs and the level of support they require is often greater than other illnesses. IHNC symptoms cause major changes to basic functions, such as: being unable to talk; severe swallowing problems with a high choking risk; breathing difficulties requiring a hole in the neck (tracheostomy). The manner of death can be highly traumatic and frightening e.g. catastrophic bleeding from the neck. Despite this poor outlook, little is known about patients' needs in the last year of life. However, IHNC patients have more emergency hospital visits compared with other cancer groups. Patients from poorer areas are more likely to die in hospital. Furthermore, head and neck cancer (HNC) units are centralised, with access to specialist services dependent on where the patient lives.

The researcher wishes to understand 'stress points' in the patients' journey, where things do not go as planned, identify priorities for change and develop patient-led solutions.

There are two main parts to this work, occurring over 21-months across Yorkshire, Northwest and Northeast England.

1. A series of up to three interviews with approximately 25 IHNC patients and their families, along with group discussions with healthcare workers involved in IHNC care. These will explore how patients' needs and use of healthcare change over time.
2. Using interview and group discussion findings, the study team will hold a series of workshops with patients, families, clinical service leaders, and healthcare workers. The study team will identify priorities and develop ways to improve care experiences.

The research is funded by the National Institute for Health Research (NIHR) Research for Patient Benefit programme.

DETAILED DESCRIPTION:
STUDY DESIGN - A prospective longitudinal qualitative study across three regions of North England, accompanied by co-design workshops which will utilise study findings to identify priority areas for improving care for patients with incurable Head and Neck Cancer (HNC).

SETTING - Three HNC centres based in Northwest, Northeast and Yorkshire representing areas of high incidence of HNC, diverse socioeconomic populations and heterogenous geographical locations (main sites - Newcastle Upon Tyne Hospitals National Health Service (NHS) Foundation Trust, Liverpool University Hospitals NHS Foundation Trust and Sheffield Teaching Hospitals NHS Foundation Trust).

METHODS

Work package 1: Longitudinal qualitative study (months 1-18) This will comprise of longitudinal interviews with patients and family carers (WP1a) and focus groups with healthcare professionals (WP1b).

WP1a: Longitudinal interviews Rationale for study design: Previous qualitative HNC studies all entailed participants being asked once about their experiences. Longitudinal interviews shed light on how issues evolve over time and are particularly suitable when there is an unpredictable disease trajectory; changing needs; and interactions with healthcare services are varied and complex. They offer advantages over a single interview or a comparison of 'snapshot' data at different stages in an illness. These include: capturing change over time; facilitating more private, evolving accounts; and exploring how external factors, such as the influence of healthcare services over the course of the patient journey, affect needs and experiences. They can highlight shortcomings and allow suggestions for improvements. Additionally, longitudinal interviews facilitate a continuing relationship between the researcher and participant bringing personal satisfaction to both parties as well as helping make any 'after-death' interviews with family carers more acceptable. The feasibility and acceptability of longitudinal interviews with people with incurable disease are demonstrated by Murray et al (2009). They report on longitudinal interviews conducted with more than 150 palliative care patients (including those with lung cancer, brain tumours, severe chronic obstructive airways disease and advance cardiac failure).

Study population: Incurable HNC patients and/or their family carer.

Sampling: The study team will recruit a range (n=18-25) of HNC patients (+/- their family carer) over an initial 7-months (aiming to conduct up to 60 interviews). Maximum variety sampling will be undertaken using variables anticipated to experience differences in care and outcomes e.g. age, gender, ethnicity, living alone, and postcode (to determine distance from cancer centre and link to Index of Multiple Deprivation). A matrix will be constructed with the selected variables and will be reviewed after each participant is recruited to determine which groups have been 'captured' and to target further recruitment to where 'gaps' exist. Liaison with clinical colleagues to highlight these 'gaps' will help direct ongoing recruitment.

Recruitment: Potential participants will be identified through HNC and Specialist Palliative Care Multi-disciplinary Team (MDT) meetings, outpatient clinics (both face-to-face and virtual consultations), in-patient and community settings. Initial approaches via local healthcare professionals will be tailored to each site.

Data collection: Participants will be invited to take part in 3 qualitative, semi-structured interviews at 4 monthly intervals. Interviews (video, telephone or if limited verbal communication, face-to-face or online written interviews) will be conducted depending on COVID restrictions/participant preferences at a time and place of their choice. Online written interviews use a shared document e.g., Google Docs, during the online interview and enable the interview to be conducted in writing (if a potential participant is unable to verbalise). Both the interviewer and interviewee will have access to the shared document. Initially, an introductory paragraph from the topic guide will be pasted into the online shared document by the interviewer. The interviewer will then type in the first question and allow the interviewee to type their response.

The interview length will be determined by the patients' ability to participate, aiming for approximately 45 minutes. Subsequent interviews will be approximately 30 minutes and more focused on changes since the last interview. Interviews will be open and conversational loosely following the topic guide (developed in collaboration with PPI group), using a blended approach of interview techniques, with passive interviewing allowing the participant space and time to tell their story (narrative), and more active techniques, including appreciative inquiry employed. Interviews will be digitally recorded, with the participants' consent, with field notes made to include any additional comments or reflections by the researcher.

Baseline demographic data will be collected from the participant and will include age, gender, ethnicity, postcode, and whether or not they live alone. Key clinical information (collected via a standard form) will be obtained directly from clinical teams or from the hospital records via members of the research team. The information will include date of diagnosis, type of head and neck cancer, whether localised or metastatic disease, reason for incurability of head and neck cancer.

With consent, and if preferred, patients will be asked if they wish to nominate a family carer, either to support the interview process and participate in a joint interview (representing a 'unit of care'); or to participate in an interview themselves if the patient was unable to do so. The study team will sensitively discuss the uncertainty about the future and the possibility, that if the patient became too unwell (or died), advanced consent can be given for their family carer to be interviewed in their absence. This approach has been used previously by the applicant team in palliative care studies (Mayland). For patients who become too unwell (or die) during the course of the study, their family carer will be approached to discuss whether they wish to participate in a further interview.

Analysis: The interviews will be digitally recorded, transcribed verbatim by a recommended University transcription service, and the transcripts will be anonymised. Analysis will be supported using NVivo (qualitative data analysis software) and conducted using a framework approach. Framework analysis facilitates both rigorous, transparent data management but enables analysis to move backwards and forwards without losing sight of the 'raw' data. The five stages are: familiarisation; identification of the thematic framework; indexing; charting; and mapping and interpretation. The framework will be developed from the principles of Picker's 'Patient Centred Care' but may include areas beyond this to account for additional issues identified.

WP1b: On-line focus groups with healthcare professionals (HCP) (Months 13 & 14) Rationale: Focus groups represent a type of group interview, bringing benefit from the communication and interaction between research participants. Generally, they involve 6-10 people, and as multidisciplinary teams are involved in HNC care, represent an effective way to seek views about our research aims compared with conducting individual interviews. Through the COVID-19 pandemic, online methods of group discussion have become more viable and offer advantages including: widening participation across larger geographical areas; being more time-efficient for clinical staff; and reducing costs compared with face-to-face meetings. However, it can be more challenging to manage discussions and ensure engagement in online focus groups and it has been recommended to include no more than five participants.

Study population: Healthcare professionals involved in the case of incurable HNC patients over the last 12 months

Sampling: The study team aim to involve approximately 20 HCP. Up to 5 focus groups will be conducted, each involving approximately 5 people. A purposive, snowball sampling strategy will be used to gain views from different HCP perspectives, working within the Northwest, Northeast and Yorkshire. The sample will be stratified to seek representatives from the following groups: HNC multidisciplinary team member (surgeon, oncologist, Clinical Nurse Specialist, allied health professionals); specialist palliative care (SPC); and primary and community care (General Practitioners and District Nursing).

Recruitment: HCPs will be identified utilising a variety of different forums including:

* Newly established NIHR partnership project - PP-HANC network (which links the Clinical Research Network areas of the North East and North Cumbria, Northwest Coast and Yorkshire and Humber) including via social media.
* Regional HNC MDT meetings
* SPC MDT meetings
* Bulletins and email dissemination (within primary care and hospital trusts), existing networks, and social media.

Within these forums, the contact details for the research team and the Participant Information Sheet will be disseminated. Interested, eligible people will be invited to contact the research team. Alternatively, with verbal consent, their contact details can be forwarded to the research team via one of the study's collaborators.

Data collection: The focus groups will be conducted on-line, via a University of Sheffield approved video-conferencing system and recorded. The focus group sessions will last up to 90 minutes and loosely follow a topic guide.

Analysis: With consent, the focus groups will be digitally recorded, and field notes taken. The focus groups will be transcribed verbatim by a recommended University transcription service, and the transcripts will be anonymised. Analysis will be supported using NVivo and will use a similar framework to the patient interviews, being mindful of any new factors discussed not previously mentioned by patients and family carers. Any identifiable data will be removed from the analysis. Pattern-matching across the patient and HCP coding matrix will identify areas of congruence and incongruence.

Work package 2: Co-design workshops (months 18-20) Design: The study team will follow the co-design approach of O'Brien and colleagues to integrate scientific evidence, expert knowledge and experience, and stakeholder involvement to start the process of prioritising and developing innovative solutions and interventions to help improve experiences with healthcare services for those with incurable HNC. A hybrid approach will be used incorporating initial 'virtual' information exchange meetings lasting approximately 60 minutes. Then, two face-to-face co-design workshops (unless these need adaptations due to COVID restrictions) will be conducted, lasting approximately 3 hours.

Outcomes: Initial logic model; list of innovative solutions; decision about priority areas for intervention development.

Stakeholders: Approximately 15 stakeholders as well as project team members and three PPI representatives from our existing group.

Individuals with 'lived experience' (n=5-8). In addition to three PPI representatives, the study team will involve HNC patients and those who have been involved in caring for someone with HNC (family and friends). They will be approached using a variety of routes including current study participants, existing contacts through HNC support groups and charities (e.g., Swallows), our NIHR Partnership project (PP-HANC), and our HCP co-leads (Mayland, Patterson) and clinical colleagues. Healthcare professionals, commissioners and service leads (n=5-8). The study team will include a diverse group and approach HCP, commissioners, and service leads involved in the funding and provision of care for incurable HNC patients. Healthcare professionals who work within the community (GPs, community nurses, SPC professionals) and hospital setting (oncologists, allied health professionals, clinical nurse specialists) will be considered. In addition to the approaches listed above, stakeholders will be contacted through current linkages with our NIHR Partnership project (PP-HANC), Cancer Alliances, the emerging Integrated Care Systems, and partnerships such as the Liverpool Head and Neck Centre.

Methods Invitation: Those interested will be approached using both verbal and written means. With permission, they will be contacted by the researcher to have the opportunity to ask questions/have further discussions. Consent will be obtained for participation in the three co-design workshops. If the participant wishes to proceed, they will be sent a link to an online consent form. Prior to first workshop, the research team will confirm the participant has read the Participant Information Sheet and completed the online consent form. If the consent form has not been received by the time of the initial meeting, recorded verbal consent will be obtained. A copy of the agreed consent form will be sent to the participant and the verbal recording of consent will be stored separately to the main interview recording. Permission to audio-record the meetings and co-design workshops will be obtained. These will not be transcribed but will form an additional account of the workshops.

Initial information exchange meetings (month 18) Purpose: To build relationships and present an overview of the study; provide opportunity for participants to share their experiences and how they relate to the preliminary study findings; outline the purpose of the co-design workshops.

Setting: The initial information exchange meetings will be held online.

Outcomes: Key stakeholders informed about subsequent co-design workshops; increased awareness of local contextual differences and lived experiences.

Methods: Two group meetings will be conducted virtually - one for those with lived experience and one for other stakeholders. By having initial meetings in a smaller format, this supports the sharing of lived experiences, local contextual differences and enables these to influence and shape the subsequent iterative work. A summary of our preliminary qualitative interview and focus group findings will be presented and details about the processes used in subsequent workshops.

Co-design workshop 1 (month 19) Purpose: To identify and prioritise 'stress-points' in the system, where things need to be improved, and generate initial ideas for solutions.

Outcomes: Collation of workshop ideas to help identify the initial elements of a preliminary logic model.

Setting: The workshop will take place in-person in a location accessible to all stakeholders.

Methods: Prior to the workshops, the study team will generate a series of vignettes from our interview findings that stakeholders can engage with to stimulate discussion. The vignettes will represent personas (representing a different HNC patient) with specific characteristics, circumstances and challenges reflecting real life experiences relating to healthcare service use that arose from the interviews and focus groups. The vignettes will be informed by PPI engagement (month 16), clinical experiences and our systematic reviews. Within the co-design workshop, discussion about the vignettes will be based around the principles of 'Patient Centered Care' and how well or not each of these are addressed. Stakeholders will work collaboratively and iteratively to discuss key issues and the potential reasoning. Ideas will be generated about what would be useful and/or needed to achieve patient-centered care and experience. The research team have excellent facilitation and communication skills to ensure all voices are heard. Following the workshop, the research team will use the ideas and discussion, to begin the process of identifying the initial elements of a logic model (contextual issues, mechanism, outcomes) mapping the issues across the incurable HNC patient journey.

Co-design workshop 2 (month 20) Purpose: To present initial elements of a logic model; To generate potential solutions and consider interventions in the context of barriers, facilitators, strengths and weaknesses

Outcome: List of potential solutions and priority areas for intervention development; Refined logic model

Setting: The workshop will take place in-person in a location accessible to all stakeholders.

Methods: Key stakeholders will be provided with the ideas about potential solutions and the initial elements of a logic model. Using the principles of the 'Six Hats Exercise', participants will be invited to discuss the barriers, facilitators, strengths and weaknesses from different perspectives (i.e. each 'hat' will represent different people, such as a person with HNC, family member, oncologist to help consider other viewpoints). Further discussion will draw together priority areas for intervention development and the elements of a refined logic model (resources, activities, contextual issues, mechanisms, outputs and outcomes).

Next steps: Following the co-design workshops, the research team will bring together the findings into a refined logic model and the potential areas for future intervention development (in keeping with the Medical Research Council guidance). This will inform a follow-on grant application, seeking to develop, optimize and conduct initial feasibility testing for an intervention to improve experiences for those with incurable HNC and their families.

ELIGIBILITY:
Inclusion Criteria:

* INTERVIEWS WITH PATIENTS AND CARERS

  * Have a clinical diagnosis of incurable HNC where the intent of any treatment is palliative, including those with:

    * incurable primary HNC
    * recurrent or persistent HNC not amenable for further curative treatment
    * metastatic disease
    * other co-morbidities (including a concurrent primary cancer at another site) meaning curative treatment is either not advised by the MDT or reflected by the patients' choice
  * Are >= 18 years old
  * Able to give informed consent
  * Reside within the networks covered by the three chosen HNC centres
  * Or are/was a family carer (>= 18 years old) to someone participating in the study.

FOCUS GROUPS WITH HEALTHCARE PROFESSIONALS

* Any HCP who has been involved in the case of incurable HNC patients over the last 12 months
* Works clinically within the regions of the Northwest, Northeast or Yorkshire (in keeping with the Clinical Research Network areas of the North East and North Cumbria, Northwest Coast and Yorkshire and Humber https://local.nihr.ac.uk/lcrn/).
* Are >= 18 years old
* Able to give informed consent
* Able to participate in an online focus group, when required.

Exclusion Criteria:

* INTERVIEWS WITH PATIENTS AND CARERS

  * Unable to provide fully informed written consent FOCUS GROUPS WITH HEALTHCARE PROFESSIONALS
  * Unable to provide informed consent
  * Unable to participate in an online focus group, when required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Head and Neck Cancer and their carers/ family. Healthcare Professionals
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Completion of interviews in Work Package 1a | Within 18 months of consent
  Completion of interviews in Work Package 1a
Completion of on-line focus groups in Work Package 1b | Within 12 months of being involved in the care of HNC patients
  Completion of interviews in Work Package 1a
Completion of co-design workshops in Work Package 2 | Within 20 months of consent
  Completion of co-design workshops in Work Package 2

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Mayland, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided